CLINICAL TRIAL: NCT04763993
Title: Reflux Disease After Gastric Bypass Versus Sleeve Gastrectomy in Morbid Obese Patients: an Italian Monocentric Randomized Clinical Study (ReBvSS)
Brief Title: Reflux Disease After Gastric Bypass Versus Sleeve Gastrectomy in Morbid Obese Patients: an Italian Study
Acronym: ReBvSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ReBvSS
Record Dates: First submitted 2021-02-10; First posted 2021-02-21 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Gastroesophageal Reflux Disease; Obesity
Keywords: Gastroesophageal Reflux Disease; Obesity; Sleeve gastrectomy; Gastric bypass; DeMeester score; pH-monitoring
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RYGBP (Active Comparator): RYGBP: Roun-en-Y Gastric Bypass
  Interventions: Procedure: Roux-en-Y-Gastric bypass, Sleeve gastrectomy; Procedure: SG
- SG (Experimental): SG: Sleeve Gastrectomy
  Interventions: Procedure: Roux-en-Y-Gastric bypass, Sleeve gastrectomy; Procedure: SG

INTERVENTIONS:
Procedure: Roux-en-Y-Gastric bypass, Sleeve gastrectomy — RYGBP consists in creating a small gastric pouch along the little curvature of the stomach, followed by the section of the small bowel. The restoration of the gastro-intestinal tract is achieved by performing a gastro-jejunal and a jejuno-jejunal anastomosis, giving this procedure the characteristic aspect of a Y. Also, for RYGBP the laparoscopic approach requires the placement of 5 trocars in the upper part of the abdomen.
Procedure: SG — SG consists in removing the fundus and the body of the stomach, along the greater curvature. To perform it with a laparoscopic approach, we create the pneumoperitoneum with Veress needle and place 5 trocars in the upper part of the abdomen. The first step is the dissection of the greater curvature of the stomach, that starts at 6 centimetres from pylorus and it's conducted up to the angle of His, freeing the fundus and exposing the left pillar. A 38 Fr bougie is placed inside the stomach to calibrate its section. After it is carried out, the specimen is removed from the greater trocar site.

SUMMARY:
The study aims to clarify if GERD, defined by results of 24 hours potential of hydrogen (pH) monitoring and abnormal DeMeester Score (DMS), in obese patients could worsen after Sleeve Gastrectomy (SG) more than after RYGBP. To demonstrate this hypothesis, the investigators will study the obese population suspected for GERD with 24 hours monitoring and High-Resolution Esophageal Manometry (HRM). DMS is calculated pre-operatively and, once GERD is confirmed, the patients are enrolled for randomization to SG or RYGBP. The suspicion of GERD is investigated with the GERDQ score and EGDS, that all obese patients have pre-operatory.

DETAILED DESCRIPTION:
Obesity is an independent risk factor for GERD and its complications. Bariatric surgery is effective in treatment of obesity and at the same time in controlling GERD, but there is disparity in current literature if sleeve gastrectomy could worsen it, more than gastric bypass. Our study aims to investigate if there is a difference in postoperative GERD between these two surgical procedures in obese patients with pre-existing GERD, defined by results of 24 hours pH monitoring, expressed by an abnormal DeMeester Score (DMS). REBvSS is a monocentric randomized controlled trial (RCT). The investigators will study 128 obese patients, eligible for Bariatric Surgery (BMS), suspected for GERD, with 24-h pH monitoring and high-resolution manometry. DMS is calculated pre-operatively and, once GERD is confirmed, the patients are randomized to SG or RYGBP. The DMS is then calculated on 24 hours pH monitoring 24 months after the surgery and the degree of GERD is evaluated. The promoter centre is the Division of Minimally invasive Oncological General Surgery at Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan, Lombardy, that is an excellence centre for bariatric and metabolic surgery according to Società Italiana di Chirurgia dell'Obesità e delle malattie metaboliche (SICOB) accreditation policy, where the study will be carried out.

Medical history will be collected during the first outpatient examination and assessed as follows:

* Diagnosis of Obesity, based on value of BMI ≥ 35;
* Investigation of obesity-related diseases
* Clinical, nutritional and surgical history
* GERDQ score If the patient is eligible for BMS and there is the suspicion of GERD the preoperative evaluation will be carried out. It consists of a trial specific evaluation (EGDS, 24-h pH monitoring, HRM, DMS), that confirms the presence of GERD, and a standard evaluation (Ultrasonography of abdomen, ECG, Chest X-Ray, Blood exams, anesthaesiologic evaluation). When all the inclusion criteria are verified, the patient will be randomized to RYGBP or SG group and will undergo surgery. All patients will be randomized centrally using an online computer controlled permuted-block randomization module between SG and RYGBP in a 1:1 ratio.

The postoperative visits will be organised as follow:

* 90 days after surgery, to evaluate the presence or the absence of medical or surgical complications;
* 12 months and 24 months after surgery EGDS, 24 hours pH-monitoring and HRM will be performed to evaluate the degree of esophagitis and calculate the DMS; the quality of life and the symptoms will be assessed troughs BAROS and GERDQ score; also the trend of comorbidities will be examined.

Every patient will be analysed according to the allocated treatment. The investigators hope that our study will finally answer this issue, thanks to its randomized nature and the definition of GERD based on gold standard pH monitoring. These findings might influence decision-making in bariatric surgery and change or confirm the success of sleeve gastrectomy, also for what concerns the reflux disease.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance of randomization to surgery;
* Participant is willing and able to give informed consent for participation in the trial;
* Written informed consent;
* Compliance to follow-up;
* Male and female;
* ≥18 and ≤70 years old;
* BMI ≥ 35 with obesity-related comorbidities;
* BMI ≥ 40 with or without obesity-related comorbidities;
* GERDQ score ≥ 3 points;
* Use of proton pump inhibitor;
* Mild and Moderate GERD (DMS ≥14.72 ≤100)
* Incompetence of the Esophagogastric junction
* Los Angeles grade A, B, C, D esophagitis.

Exclusion criteria

* Medical or psychiatric conditions that compromises the patient's ability to give informed consent or comply with the study protocol;
* Barrett's esophagus (BE);
* Spastic motor disorders and esophageal hypomotility;
* Peptic strictures;
* Absence of GERD (DMS<14.72);
* Severe GERD (DMS>100);
* Hiatal hernia > 5 cm;
* Previous bariatric surgery or major general surgery;
* Type 2 diabetes (T2D) for more than > 5 years;
* Necessity to explore stomach, the duodenum or the biliary tract;
* Refuse of randomization;
* Personal reasons.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Change of the pre-existing Gastro-Esophageal Reflux Disease (GERD) from baseline in patients underwent SG and RYGBP | Change from baseline DeMeester Score 24 months after surgery
  GERD will be evaluated performing 24-h pH monitoring before the surgery. The presence and the degree of GERD will be quantified calculating the DeMeester Score (DMS):
  * DMS < 14.72 there is no evidence of GERD;
  * DMS 14.72 - 50 mild GERD;
  * DMS 50 - 100 moderate GERD;
  * DMS > 100 severe GERD An upgrading in DMS class will determine a worsening in GERD

SECONDARY OUTCOMES:
Postoperative Gastroesophageal Reflux Disease (GERD) from baseline | Change from baseline DeMeester Score 12 months after surgery
  The degree of GERD will be quantified calculating the DeMeester Score (DMS):
  * DMS < 14.72 there is no evidence of GERD;
  * DMS 14.72 - 50 mild GERD;
  * DMS 50 - 100 moderate GERD;
  * DMS > 100 severe GERD An upgrading in DMS class will determine a worsening in GERD
Postoperative reflux symptoms | Baseline and 12 and 24 months from the surgery
  Expressed by Gastroesophageal Reflux Disease Questionnaire (GERDQ) Scoring How many times per week do each of the following symptoms occur per week Score 0: Occurs on 0 days Score 1: Occurs on 1 day Score 2: Occurs on 2-3 days Score 3: Occurs on 4-7 days Questions (Score 0-3 for each based on above) Burning feeling behind the Breastbone (Heartburn)? Stomach contents moving up to the throat or mouth (regurgitation)? Pain in the middle of the upper Stomach area? Nausea? Trouble getting a good night's sleep because of Heartburn or regurgitation? Need for over-the-counter medicine for Heartburn or regurgitation? Examples: Tums, Rolaids, Maalox, or other Antacids) In addition to the medicine your doctor prescribed Interpretation Total score of 0-2 points Likelihood of GERD: 0 percent Total score of 3-7 points Likelihood of GERD: 50 percent Total score of 8-10 points Likelihood of GERD: 79 percent Total score of 11-18 points Likelihood of GERD: 89 percent
Quality of life Questionnaire | month 12 and 24 after surgery
  Expressed by Bariatric Analysis and Reporting Outcome System (BAROS) Score, calculated after 12 and 24 months from the surgery. The scoring key is assessed as follows: Failure ≤1 point; Fair > 1 to 3 points; Good > 3 to 5 points; Very Good > 5 to 7 points; Excellent > 7 to 9 points
Trend of the obesity-related diseases (Arterial hypertension, Type 2 Diabetes, continuous positive airway pressure (CPAP) use | month 12 and 24 after surgery
  Anti-hypertensive drugs (AH) taken before surgery:stability=no change in AH,resolution= no AH,improvement=decrease in AH,worsening=increase in AH In no hypertension pts before surgery;new onset=introduction of AH Oral anti-glycemic (AG) medication taken before surgery:Stability=no change in number of oral AG.Resolution=defined as no oral AG,Improvement=decrease in number of oral AG,Worsening=increase in number of oral AG or switch to insulin-dependence In pts with insulin dependence before surgery:Stability=no change in number of insulin units,Resolution=no anti-diabetic therapy,Improvement=decrease in number of insulin units or oral AG,Worsening=increase in number of insulin units In pts not affected by type 2 diabetes before surgery:new onset=introduction of anti-diabetic therapy In pts using CPAP before surgery:Stability=continued use of CPAP,Resolution=discontinued use of CPAP In pts not affected by obstructive sleep apnea syndrome (OSAS) before surgery:new onset=use of CPAP
Demographic | Enrollment
  Demographic data
Medical/Surgical complications | day 90
  The number of patients that experienced medical and/or surgical complications within 90 days from surgery, graded according to Clavien-Dindo classification (grade I, II, IIIa, IIIb, Iva, IVb, V)

IPD SHARING:
Plan to Share IPD: Undecided